CLINICAL TRIAL: NCT01632280
Title: "Neuroband": The Effect of Perioperative Enhancement of the Brain Circuit of Inhibitory Control in Obese Patients Undergoing Laparoscopic Adjustable Gastric Banding (LAGB)
Brief Title: Enhancement of Brain Circuit of Inhibitory Control in Obese Patients Undergoing Gastric Banding
Acronym: "Neuroband"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Miguel Alonso-Alonso, MD, Assistant Professor of Surgery, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012P000121; 5P30DK046200-20 (NIH)
Record Dates: First submitted 2012-06-20; First posted 2012-07-02 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Obesity
Keywords: Obesity; Gastric Banding; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Obesity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Active Comparator): In this arm, participants will receive active tDCS (2mA, 20 min per session). The anode electrode will be placed over the right inferior frontal gyrus, defined as F8 (10-20 EEG system), with the cathode electrode placed over the contralateral supraorbital area, above the left eyebrow. During each session they will also perform a computerized task designed to engage the inhibitory control circuit when confronted with food stimuli.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Participants will receive sham tDCS sessions with the same duration and electrode montage as in the real tDCS arm. In this case, current will be applied for 30 s only according to standard procedures, and participants will perform a control task where they will observe and provide responses for the same food and non-food pictures as in the active group task, but without requirement of inhibitory control for performance.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS is a well-established, safe and noninvasive neuromodulation technique that is based on the application of a weak direct current to the scalp that flows between two electrodes-anode and cathode. Although there is substantial shunting of current in the scalp, sufficient current penetrates the brain to modify the transmembrane neuronal potential, and thus influence the level of excitability and modulate the firing rate of individual neurons.
  In this study, participants will receive 10 daily sessions of tDCS (sham/real) over a period of two weeks.
  Other Names: Eldith Neuroconn DC Stimulator

SUMMARY:
In this project the investigators aim to improve eating control and weight loss outcomes in patients undergoing LAGB with an innovative brain-based intervention. Specifically, the investigators will enhance the activity of the right inferior frontal gyrus, a core region of the brain circuit of inhibitory control, using transcranial direct current stimulation (tDCS).

DETAILED DESCRIPTION:
Laparoscopic Adjustable Gastric Banding (LAGB) is a minimally invasive and reversible procedure in bariatric surgery that has a good safety record. Despite these advantages, success rates following LAGB are quite variable across individuals. Recent data suggest that complementing LAGB with interventions targeting factors along the brain-behavior spectrum could enhance weight loss results following this procedure.

The study will have the following three aims:

Aim #1: To evaluate whether enhancement of the right inferior frontal gyrus with tDCS in patients undergoing LAGB can improve inhibitory control capacity. For this aim the investigators will evaluate participants' performance in a computerized test of inhibitory control. Results from this aim will provide evidence for target engagement, and thus confirm that the brain circuit of interest was affected as a result of the intervention.

Aim #2: To examine whether enhancement of the right inferior frontal gyrus with tDCS in patients undergoing LAGB can lead to improvements in a self-reported measure of eating control (disinhibition subscale of the three-factor eating questionnaire). Results form this aim will provide evidence for an effect of the intervention on an intermediate, behavioral variable.

Aim #3: To preliminary evaluate whether enhancement of the right inferior frontal gyrus with tDCS in patients undergoing LAGB can improve postoperative weight loss outcomes. This aim will provide preliminary evidence for the clinical efficacy of the intervention over a time window period of 12 months. Weight loss at 12 months will be the primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-55 years old
* BMI: 35-60 kg/m2
* Planning to undergo or having undergone laparoscopic adjustable gastric banding (LAGB) within the previous week

Exclusion Criteria:

* Unstable medical conditions including poorly controlled diabetes and hypertension
* Pregnancy or planning pregnancy during study period
* Personal or family history of epilepsy or other unexplained loss of consciousness
* Current or past medical history of skin disease or damaged skin on the scalp at site of stimulation
* Active psychiatric or neurological condition
* Prior neurological procedure
* Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculoperitoneal shunt
* Intake of common medications that affect the central nervous system will be allowed if determined okay by MD

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12-31 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Alonso-Alonso, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Bueter M, Thalheimer A, Lager C, Schowalter M, Illert B, Fein M. Who benefits from gastric banding? Obes Surg. 2007 Dec;17(12):1608-13. doi: 10.1007/s11695-007-9263-3. Epub 2007 Nov 21. PMID 18030543
- [Background] Chevallier JM, Paita M, Rodde-Dunet MH, Marty M, Nogues F, Slim K, Basdevant A. Predictive factors of outcome after gastric banding: a nationwide survey on the role of center activity and patients' behavior. Ann Surg. 2007 Dec;246(6):1034-9. doi: 10.1097/SLA.0b013e31813e8a56. PMID 18043107
- [Background] Thalheimer A, Bueter M, Wierlemann A, Lager C, Jurowich C, Germer CT, Fein M. Predictability of outcome in laparoscopic gastric banding. Obes Facts. 2009;2 Suppl 1(Suppl 1):27-30. doi: 10.1159/000198246. Epub 2009 Mar 18. PMID 20124774
- [Background] Spitznagel MB, Garcia S, Miller LA, Strain G, Devlin M, Wing R, Cohen R, Paul R, Crosby R, Mitchell JE, Gunstad J. Cognitive function predicts weight loss after bariatric surgery. Surg Obes Relat Dis. 2013 May-Jun;9(3):453-9. doi: 10.1016/j.soard.2011.10.008. Epub 2011 Oct 29. PMID 22133580
- [Background] Bruce JM, Hancock L, Bruce A, Lepping RJ, Martin L, Lundgren JD, Malley S, Holsen LM, Savage CR. Changes in brain activation to food pictures after adjustable gastric banding. Surg Obes Relat Dis. 2012 Sep-Oct;8(5):602-8. doi: 10.1016/j.soard.2011.07.006. Epub 2011 Jul 27. PMID 21996599
- [Background] Chambers CD, Garavan H, Bellgrove MA. Insights into the neural basis of response inhibition from cognitive and clinical neuroscience. Neurosci Biobehav Rev. 2009 May;33(5):631-46. doi: 10.1016/j.neubiorev.2008.08.016. Epub 2008 Sep 11. PMID 18835296
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Aron AR, Poldrack RA. The cognitive neuroscience of response inhibition: relevance for genetic research in attention-deficit/hyperactivity disorder. Biol Psychiatry. 2005 Jun 1;57(11):1285-92. doi: 10.1016/j.biopsych.2004.10.026. Epub 2004 Dec 23. PMID 15950000
- [Background] Nitsche MA, Paulus W. Transcranial direct current stimulation--update 2011. Restor Neurol Neurosci. 2011;29(6):463-92. doi: 10.3233/RNN-2011-0618. PMID 22085959
- [Background] Goldman RL, Borckardt JJ, Frohman HA, O'Neil PM, Madan A, Campbell LK, Budak A, George MS. Prefrontal cortex transcranial direct current stimulation (tDCS) temporarily reduces food cravings and increases the self-reported ability to resist food in adults with frequent food craving. Appetite. 2011 Jun;56(3):741-6. doi: 10.1016/j.appet.2011.02.013. Epub 2011 Feb 23. PMID 21352881
- [Background] Fregni F, Orsati F, Pedrosa W, Fecteau S, Tome FA, Nitsche MA, Mecca T, Macedo EC, Pascual-Leone A, Boggio PS. Transcranial direct current stimulation of the prefrontal cortex modulates the desire for specific foods. Appetite. 2008 Jul;51(1):34-41. doi: 10.1016/j.appet.2007.09.016. Epub 2007 Dec 23. PMID 18243412
- [Background] Nederkoorn C, Houben K, Hofmann W, Roefs A, Jansen A. Control yourself or just eat what you like? Weight gain over a year is predicted by an interactive effect of response inhibition and implicit preference for snack foods. Health Psychol. 2010 Jul;29(4):389-93. doi: 10.1037/a0019921. PMID 20658826
- [Background] Nederkoorn C, Jansen E, Mulkens S, Jansen A. Impulsivity predicts treatment outcome in obese children. Behav Res Ther. 2007 May;45(5):1071-5. doi: 10.1016/j.brat.2006.05.009. Epub 2006 Jul 7. PMID 16828053
- [Background] Houben K. Overcoming the urge to splurge: influencing eating behavior by manipulating inhibitory control. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):384-8. doi: 10.1016/j.jbtep.2011.02.008. Epub 2011 Feb 24. PMID 21450264
- [Background] Batterink L, Yokum S, Stice E. Body mass correlates inversely with inhibitory control in response to food among adolescent girls: an fMRI study. Neuroimage. 2010 Oct 1;52(4):1696-703. doi: 10.1016/j.neuroimage.2010.05.059. Epub 2010 May 25. PMID 20510377
- [Background] Jacobson L, Javitt DC, Lavidor M. Activation of inhibition: diminishing impulsive behavior by direct current stimulation over the inferior frontal gyrus. J Cogn Neurosci. 2011 Nov;23(11):3380-7. doi: 10.1162/jocn_a_00020. Epub 2011 Mar 31. PMID 21452949
- [Background] Alonso-Alonso M. Translating tDCS into the field of obesity: mechanism-driven approaches. Front Hum Neurosci. 2013 Aug 27;7:512. doi: 10.3389/fnhum.2013.00512. eCollection 2013. PMID 23986687
- [Background] Kekic M, McClelland J, Campbell I, Nestler S, Rubia K, David AS, Schmidt U. The effects of prefrontal cortex transcranial direct current stimulation (tDCS) on food craving and temporal discounting in women with frequent food cravings. Appetite. 2014 Jul;78:55-62. doi: 10.1016/j.appet.2014.03.010. Epub 2014 Mar 20. PMID 24656950
- [Background] Jauch-Chara K, Kistenmacher A, Herzog N, Schwarz M, Schweiger U, Oltmanns KM. Repetitive electric brain stimulation reduces food intake in humans. Am J Clin Nutr. 2014 Oct;100(4):1003-9. doi: 10.3945/ajcn.113.075481. Epub 2014 Aug 6. PMID 25099550
- [Background] Lapenta OM, Sierve KD, de Macedo EC, Fregni F, Boggio PS. Transcranial direct current stimulation modulates ERP-indexed inhibitory control and reduces food consumption. Appetite. 2014 Dec;83:42-48. doi: 10.1016/j.appet.2014.08.005. Epub 2014 Aug 13. PMID 25128836
- See also: Beth Israel Deaconess Medical Center Website — http://www.bidmc.org
- See also: The Obesity Society Website — http://www.obesity.org
- See also: American Society for Metabolic and Bariatric Surgery Website — http://www.ASMBS.org
- See also: Weight Loss Surgery website at Beth Israel Deaconess Medical Center, Boston MA Phone 617-667-2845 — http://www.bidmc.org/wls

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between June 2012 and July 2014 from the Weight Loss Surgery Center at Beth Israel Deaconess Medical Center.
Pre-assignment Details: 2 participants withdrew from the study after enrollment but prior to assignment to a treatment arm.
Groups:
- Active tDCS: In this arm, participants received 10 daily sessions of active Transcranial Direct Current Stimulation (2mA, 20 min per session) over the course of two weeks. The anode electrode was placed over the right inferior frontal gyrus, defined as F8 (10-20 EEG system), with the cathode electrode placed over the contralateral supraorbital area, above the left eyebrow. During each session participants performed a computerized task designed to engage the inhibitory control circuit when confronted with food stimuli.
- Sham tDCS: In this arm, participants received 10 daily sessions of sham Transcranial Direct Current Sitmulation with the same duration and electrode montage as in the real tDCS arm (20 minutes, targeting the right inferior frontal gyrus). In this case, current was applied for 30 s only according to standard procedures, and participants performed a control task during which they observed and provided responses for the same food and non-food pictures as in the active group task, but without the requirement of inhibitory control for performance.
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (8.0) | 44.3 (7.1) | 43.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Participants will be weighed at the indicated time points. Weight loss at 12 months will be the primary outcome of the study.
Time Frame: Baseline, 2 weeks after surgery, 10 days of tDCS, 1 month, 3 months, 6 months and 12 months follow up
Population: 1 Participant withdrew prior to obtaining outcome data at the 10th day of tDCS, 1 participant was lost to follow-up prior to the 3-month follow-up visit, and 1 participants were lost to follow-up prior to obtaining outcome data at the 6-month follow-up visit.
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 6 | 6
pounds (lbs)
  Baseline | 285.0 (63.8) | 245.3 (41.0)
  2 weeks post gastric band (LAGB) surgery | 273.4 (62.7) | 228.4 (34.8)
  10th day of tDCS: number analyzed (Participants) | 5 | 6
  10th day of tDCS | 280.4 (62.1) | 225.8 (34.0)
  1 month follow-up: number analyzed (Participants) | 5 | 6
  1 month follow-up | 273.4 (57.0) | 220.3 (34.1)
  3 month follow-up: number analyzed (Participants) | 5 | 5
  3 month follow-up | 268 (52.1) | 210.6 (34.9)
  6 month follow-up: number analyzed (Participants) | 4 | 5
  6 month follow-up | 278.05 (52.5) | 206.5 (31.0)
  12 month follow-up: number analyzed (Participants) | 4 | 5
  12 month follow-up | 289.8 (58.8) | 204.2 (30.5)

2. Secondary Outcome: Eating Disinhibition as Measured by the Three Factor Eating Questionnaire (TFEQ)
Description: Eating Disinhibition is an eating behavior trait that reflects a tendency towards overeating and eating opportunistically in an obesogenic environment. Examples include eating in response to negative affect, overeating when others are eating, not being able to resist temptations to eat, and overeating in response to the palatability of food (Bryant, King and Blundell. Obes Rev. 2008;9:409-19). Eating disinhibition was measured using the Three Factor Eating Questionnaire (TFEQ), which contains 16 questions for this factor. Responses are scored 0 or 1 and summed, thus eating disinhibition score ranges from 0 to 16. Higher scores denote higher levels of eating disinhibition.
Time Frame: Baseline and 12 months follow up
Population: 1 participant withdrew prior to the 12 month follow-up and 2 participants were lost to follow-up prior to the 12 month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 6 | 6
units on a scale
  Baseline | 7.0 (5.4) | 3.8 (2.1)
  12 month follow-up: number analyzed (Participants) | 4 | 5
  12 month follow-up | 5.0 (1.2) | 3.6 (4.2)

3. Secondary Outcome: Change From Baseline in Inhibitory Control Over Food as Measured by the Stop Signal Reaction Task
Description: Inhibitory control over food was measured with a Stop Signal Task that was modified with the presence of distractors of two types: images of food and neutral images (control). The Stop Signal Task is a computerized task that evaluates an individual's ability to interrupt a motor response after its initiation (Logan 1994). Subjects were asked to press a response key matching the direction of an arrow, but refrain from pressing when an auditory cue ("stop signal") appeared (25% trials). The main outcome of the task is the Stop-Signal-Reaction-Time (SSRT), in milliseconds, which reflects how long it takes to inhibit a response when a stop signal appears. The SSRT is considered a laboratory measure of inhibitory control capacity. Shorter SSRT reflects more efficient inhibitory control. Here a reduction of SSRT from baseline to 12 months indicates improvement in inhibitory capacity. We provide SSRT changes for food and neutral images, reflecting specific and general effects, respectively.
Time Frame: 12 month follow-up vs. Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 4 | 5
milliseconds (ms)
  Change, stop signal reaction time, food images | -72.6 (68.3) | -51.1 (49.8)
  Change, stop signal reaction time, neutral images | -62.3 (77.8) | -46.4 (67.7)

ADVERSE EVENTS:
Time Frame: Two weeks
Description: Information about adverse events were collected using a side effects questionnaire administered at the beginning and end of transcranial direct current stimulation sessions.
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS (N=6) | Sham tDCS (N=6)
Headache (Investigations) | 1 | 2
Neck pain (Investigations) | 0 | 1
Sensations: burning, itching, or tingling (Investigations) | 1 | 3
Skin redness (Investigations) | 4 | 1
Sleepiness (Investigations) | 6 | 6
Trouble concentrating (Investigations) | 1 | 2
Acute mood change (Investigations) | 1 | 1
Warmth at the site of the electrode (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
Recruitment of participants was incomplete due to a decrease/discontinuation of gastric banding procedures throughout the duration of the study and limited funding. Findings may have also been influenced by the effect of band refills.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No